CLINICAL TRIAL: NCT02814279
Title: Evaluation of Two Different Flaps Associated With Connective Tissue Graft in the Treatment of Gingival Recession: A Randomized Clinical Trial
Brief Title: Comparison of Two Flaps for Root Coverage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, Assistant Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UEPJMF 3
Record Dates: First submitted 2016-06-23; First posted 2016-06-27 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-04

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession | interventions — Drug Prescriptions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAF plus connective tissue graft (Active Comparator): CAF treatment was performed by starting with two divergent releasing incisions lateral to the recessed area. A sulcular incision was made to unite the releasing incisions and the flap was raised beyond the mucogingival junction (MGJ) in split-full-split thickness. The connective tissue graft was removed from the palate according to Bruno technique (1994) and sutured in position. Sling sutures were placed to stabilize the flap in a coronal position 2 mm above the CEJ, followed by interrupted sutures to close the releasing incisions.
  Interventions: Procedure: CAF plus connective tissue graft; Drug: Sodium dipyrone; Drug: chlorhexidine rinse
- Tunnel plus connective tissue graft (Experimental): The tunnel flap was performed according to Zuhr et al., 2007. Following initial sulcular incisions, spit thickness flap was prepared using specific tunneling knives beyond the mucogingival junction and until flap gain mobility. The flap was laterally extended to adjacent papillae that were carefully detached by means of a full-thickness preparation. The connective tissue graft was insert into the tunnel. Sling sutures were performed involving the flap and graft to coronally cover 2 mm above the CEJ.
  Interventions: Procedure: Tunnel plus connective tissue graft; Drug: Sodium dipyrone; Drug: chlorhexidine rinse

INTERVENTIONS:
Procedure: CAF plus connective tissue graft — Periodontal surgery for root coverage by the trapezoidal flap associated with connective tissue graft.
  Other Names: Periodontal plastic surgery
  Arms: CAF plus connective tissue graft
Procedure: Tunnel plus connective tissue graft — Periodontal surgery for root coverage by the tunnel flap associated with connective tissue graft.
  Other Names: Periodontal plastic surgery
  Arms: Tunnel plus connective tissue graft
Drug: Sodium dipyrone — All participants were instructed to take 500 mg sodium dipyrone just in case of pain.
  Other Names: Drug prescription
Drug: chlorhexidine rinse — All participants were instructed to perform 0.12% chlorhexidine rinse after the surgical procedures.
  Other Names: Drug prescription

SUMMARY:
The aim of this study was to compare clinical, esthetic and patient-centered outcomes of coronally advanced tunnel (TUN) and coronally advanced flap (CAF) both associated with connective tissue graft (CTG) in the treatment of gingival recession.

DETAILED DESCRIPTION:
This is a prospective, parallel and controlled clinical trial. The population evaluated in the study was selected at Institute of Science and Technology (ICT), São José dos Campos, College of Dentistry.

Patients were assigned to one of the three treatment groups:

* Group TUN+CTG (21): Periodontal surgery for root coverage through tunnel flap technique plus connective tissue graft.
* Group CAF+CTG (21): Periodontal surgery for root coverage through trapezoidal flap plus connective tissue graft.

All surgical procedures were performed by a single operator (MPS). The gingival recession defects were randomly treated by either the trapezoidal-type of coronally advanced flap plus connective tissue graft (CAF+CTG) or the coronally advanced tunnel technique with subepithelial connective tissue graft (TUN+CTG). In brief description, CAF treatment was performed by starting with two divergent releasing incisions lateral to the recessed area. A sulcular incision was made to unite the releasing incisions and the flap was raised beyond the mucogingival junction (MGJ) in split-full-split thickness. The connective tissue graft was removed from the palate and sutured in position. Sling sutures were placed to stabilize the flap in a coronal position 2 mm above the cement-enamel junction (CEJ), followed by interrupted sutures to close the releasing incisions. The tunnel flap was performed with initial sulcular incisions, spit thickness flap was prepared using specific tunneling knives beyond the mucogingival junction and until flap gain mobility. The flap was laterally extended to adjacent papillae that were carefully detached by means of a full-thickness preparation. The connective tissue graft was insert into the tunnel. Sling sutures were performed involving the flap and graft to coronally cover 2 mm above the CEJ. After the surgery, the participants were requested to take 500 mg of sodium dipyrone every 4 hours for 3 days in case of pain, and to avoid brushing and flossing in the treated area for a period of 2 weeks. During this period, plaque control was performed using 0.12% chlorhexidine rinse used twice a day. The sutures were removed after 7 days, and all of the patients were recalled for prophylaxis and reinforcement of motivation and instruction for atraumatic tooth brushing during the study period.

Clinical, esthetics, and comfort of patients parameters were assessed at 45 days, 2, 3 and 6 months after the procedure.

Quantitative data were recorded as mean ± standard deviation (SD), and normality was tested using Shapiro-Wilk tests. The probing depth (PD), relative gingival recession (RGR), clinical attachment level (CAL), keratinized tissue thickness (KTT), keratinized tissue width (KTW), and dentin hypersensitivity (DH) values were examined by two-way repeated measures ANOVA to evaluate the differences within and between groups, followed by a Tukey test for multiple comparisons when the Shapiro-Wilk p value was ≥ 0.05. Those presenting Shapiro-Wilk p values < 0.05 were analyzed using a Friedman test (for intragroup comparisons) and Mann-Whitney tests (for intergroup comparisons). Patients' esthetics and discomfort measures using visual analog scale (VAS) were analyzed by T-tests. The frequency of complete root coverage was compared using χ2 tests. Intergroup root coverage esthetic score (RES) comparisons were performed with a T-test. A significance level of 0.05 was adopted.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting Miller class I or II gingival recession in the maxillary canines or premolars
* Visible cemento-enamel junction (CEJ) with pulp vitality;
* Patients presenting no signs of active periodontal disease and full-mouth plaque and bleeding score ≤20%;
* Patients older than 18 years old; probing depth ˂3 mm in the included teeth;
* Patients who agreed to participate and signed an informed consent form.

Exclusion Criteria:

* Patients presenting systemic problems that would contraindicate the surgical procedure;
* Patients taking medications known to interfere with the wound healing process or that contraindicate the surgical procedure;
* Smokers or pregnant women;
* Patients who underwent periodontal surgery in the area of interest;
* Patients with orthodontic therapy in progress.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mauro P Santamaria, PhD, Principal Investigator — ICT-UNESP

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] de Sanctis M, Zucchelli G. Coronally advanced flap: a modified surgical approach for isolated recession-type defects: three-year results. J Clin Periodontol. 2007 Mar;34(3):262-8. doi: 10.1111/j.1600-051X.2006.01039.x. PMID 17309597
- [Background] Zuhr O, Fickl S, Wachtel H, Bolz W, Hurzeler MB. Covering of gingival recessions with a modified microsurgical tunnel technique: case report. Int J Periodontics Restorative Dent. 2007 Oct;27(5):457-63. PMID 17990442
- [Background] Bruno JF. Connective tissue graft technique assuring wide root coverage. Int J Periodontics Restorative Dent. 1994 Apr;14(2):126-37. PMID 7928129
- [Derived] Santamaria MP, Neves FLDS, Silveira CA, Mathias IF, Fernandes-Dias SB, Jardini MAN, Tatakis DN. Connective tissue graft and tunnel or trapezoidal flap for the treatment of single maxillary gingival recessions: a randomized clinical trial. J Clin Periodontol. 2017 May;44(5):540-547. doi: 10.1111/jcpe.12714. Epub 2017 Apr 12. PMID 28231619

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At clinical site
Pre-assignment Details: The study recruited 45 eligible patients. However, three patients were excluded before assignment to groups. Two recruited patients never presented for treatment and one declined to proceed.
Period: Overall Study
Arm/Group | CAF Plus Connective Tissue Graft | Tunnel Plus Connective Tissue Graft
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CAF Plus Connective Tissue Graft | Tunnel Plus Connective Tissue Graft | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.66 (8.89) | 39.71 (10.38) | 40.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 9 | 6 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 19 | 21 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 21 | 21 | 42
Gingival recession depth [Mean (Standard Deviation); unit: millimeters] | 3.2 (0.7) | 3.0 (0.6) | 3.0 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Defect Coverage
Description: Percentage mean (%) of root surface covered by the surgical treatment, measured through a periodontal probe.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of root coverage
Arm/Group | CAF Plus Connective Tissue Graft | Tunnel Plus Connective Tissue Graft
Number analyzed (Participants) | 21 | 21
percentage of root coverage | 87.2 (27.1) | 77.4 (20.4)

2. Secondary Outcome: Root Coverage Esthetic Score
Description: The Root Coverage Esthetic Scale (RES; Cairo et al. 2009) was performed by two blinded and independent examiners (CFA and IFM) at the 6-month post-operative assessment. This score evaluates five variables: level of the gingival margin, marginal tissue contour, soft tissue texture, mucogingival junction alignment, and gingival color. Because complete root coverage was the primary treatment goal, and the other variables were considered secondary, the value assigned for root coverage was 60% of the total score, whereas 40% was assigned to the other four variables. With regard to the assessment of the final position of the gingival margin, 3 points were given for partial root coverage, and 6 points were given for complete root coverage; 0 points were assigned when the final position of the gingival margin was equal or apical to the previous recession. One point was assigned for each of the other four variables. Thus, 10 points was a perfect score.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: photographs
Arm/Group | CAF Plus Connective Tissue Graft | Tunnel Plus Connective Tissue Graft
Number analyzed (Participants) | 21 | 21
Number analyzed (photographs) | 42 | 42
units on a scale | 8.12 (1.55) | 7.98 (1.74)

ADVERSE EVENTS:
Arm/Group | CAF Plus Connective Tissue Graft | Tunnel Plus Connective Tissue Graft
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No